CLINICAL TRIAL: NCT02154022
Title: Collection of Pharmacokinetic and Probe Substrate Samples From Participants With Unanticipated Response, Significant Toxicity or Concern of Future Toxicity
Brief Title: Collection of Pharmacokinetic Samples From People With Unanticipated Response, Significant Toxicity or Concern of Future Toxicity
Status: Enrolling by invitation | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 140128; 14-C-0128
Record Dates: First submitted 2014-05-31; First posted 2014-06-03 (Estimated); Last update posted 2026-01-05 (Actual); Status verified 2025-08-06

CONDITIONS: Cancer; Solid Tumors; Neoplasm
Keywords: PK; Natural History
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Participants who are currently enrolled in IRB approved NIH Intramural Research Program clinical trial

SUMMARY:
Background:

- Certain drugs - even when they are meant to help people - cause side effects. These are unwanted effects of the drug. There are many reasons why a drug might cause side effects in one person and not in another. It may be because of how much of the drug is in the person s blood at one time. Researchers want to study the blood of people having drug side effects to better understand why they happen.

Objective:

- To obtain blood samples from participants being treated with an investigational or FDA approved drug at the NIH who are having or are anticipated to have bad side effects that are thought to be due to large amount of the drug in their blood. The samples will be used to assess the cause of the side effects.

Eligibility:

- People 2 years and older who are currently enrolled in clinical trials at the NIH Intramural Research Program (IRP).

Design:

* Participants will give blood samples.

DETAILED DESCRIPTION:
Background:

* Pharmacology is the study of pharmaceutical compounds, and encompasses several parameters, including how the body handles the substance (pharmacokinetics, PK), what the substance does to the body at the molecular level (pharmacodynamics), overall efficacy (response), and any adverse events or toxicity encountered.
* The Clinical Pharmacology Program (CPP) within the Center for Cancer Research (CCR) of the National Cancer Institute (NCI) has sensitive, state of the art bioanalytical instrumentation that can accurately and precisely quantitate drug concentrations in plasma.
* Currently, the CPP can only analyze samples from clinical trials that have explicit instructions (within the Pharmacokinetics section) to do so in the IRB approved protocol.
* However, clinical trial protocols without a Pharmacokinetics section may still need occasional pharmacokinetic plasma samples drawn and drug concentration measurements performed to help explain unexpected AEs or toxicity or anticipated altered pharmacokinetics.
* The administration of probe substrates can be used to determine the phenotype of enzymes and transporters responsible for drug disposition, providing a useful tool to better understand the cause of unexpected AEs or toxicities of clinical trial participants.

Objectives:

* Primary Objective: To assess PK samples/profiles from participants being treated with an investigational agent or FDA approved therapy at the NIH who are exhibiting or are anticipated to exhibit unusual response or toxicity that is believed to be due to high drug concentration in order to assess the cause of the toxicity and adverse events.
* Exploratory Objective: To use phenotyping probes to research how individuals with genetic defects in drug metabolism genes might handle the probe, assessing blood concentrations to ascertain the rate of metabolism of enzymes and transporters.

Eligibility:

- Any participants who are currently enrolled in IRB approved NIH Intramural Research Program (IRP) clinical trials are eligible.

Design:

* The CPP will measure the drug plasma concentration (or send the sample out to a third party if the assay is commercially available).
* The CPP will measure the plasma concentration of enzyme or transporter phenotyping probe substrates (or send the sample out to a third party if the assay is commercially available) in select participants enrolled on clinical trials at the CCR.
* The accrual ceiling for this study is 100 participants. The anticipated accrual rate for this protocol is less than 10 participants per year, and based on the accrual ceiling, the duration of accrual and the total study duration is 10 years.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Any individuals greater than or equal to 2 years of age who are currently enrolled in IRB approved NIH Intramural Research Program (IRP) clinical trials are eligible. (Exception: Participants <18 years old will not be eligible for probe administration.)
* Ability of subject or a Legally Authorized Representative (LAR) to understand and the willingness to sign a written informed consent document.
* Individuals who have received or are anticipated to receive an investigational agent or FDA approved therapy at the NIH who meet one of the following criteria:

  * Individuals in whom altered pharmacokinetics are anticipated to occur based on pharmacogenetics, history of toxicities with similar agents, drug interactions, or other patient-specific factors which may alter absorption, distribution, metabolism, or excretion. OR
  * Individuals who are exhibiting unusual response or toxicity that is believed to be due to high drug concentration in order to assess the cause of toxicity and adverse events.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Any participants greater than or equal to 2 years of age who are currently enrolled in IRB approved NIH Intramural Research Program (IRP) clinical trials are eligible.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-07-31 (Actual); Primary Completion 2029-05-01 (Estimated); Study Completion 2030-05-01 (Estimated)

PRIMARY OUTCOMES:
To obtain PK sample | study completion
  Measure drug concentrations in blood.

CONTACTS AND LOCATIONS:
Overall Officials: William D Figg, Pharm.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2014-C-0128.html